CLINICAL TRIAL: NCT01777581
Title: A Ten-Week, Randomized, Double-Blind, Placebo-Controlled Parallel-Group Study of Milnacipran for Radicular Pain Associated With Lumbosacral Disk Disease
Brief Title: Milnacipran for Lumbosacral Radicular Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00020888; SAV-MD-12
Record Dates: First submitted 2012-11-30; First posted 2013-01-29 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-04

CONDITIONS: Radicular Pain Related to Lumbosacral Disc Disease
Keywords: sciatica radiculopathy lumbar disc lumbosacral disc
MeSH Terms: interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- milnacipran (Experimental): Milnacipran, flexibly dosed
  Interventions: Drug: Milnacipran
- Sugar pill (placebo) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran
  Other Names: Savella
  Arms: milnacipran
Drug: Placebo
  Arms: Sugar pill (placebo)

SUMMARY:
This study investigates whether milnacipran reduces radicular pain ("sciatica") in patients with lumbosacral disc disease.

DETAILED DESCRIPTION:
The current study evaluates the potential efficacy of milnacipran in reducing lower extremity radicular pain associated with lumbar disk disease. Milnacipran will be titrated based on efficacy and tolerability aimed at the higher end of the therapeutic range; a recent study of a serotonin norepinephrine reuptake inhibitor in patients with osteoarthritis pain suggests efficacy may be dose related. Patients are likely to have concomitant nociceptive lower back pain, and cotreatment with opioids, muscle relaxants, benzodiazepines, or nonsteroidal anti-inflammatory drugs at stable doses will be permitted. Patients participating in stable regimen of physical therapy or biofeedback will be eligible. Procedural interventions (e.g. epidural steroid injection, nerve block, facet radioablation, acupuncture) during the study and 3 months prior will be exclusionary. Anticonvulsants, tramadol, and other antidepressant drugs will be excluded.

The study is a ten-week randomized, double-blind, placebo-controlled trial (RCT) of milnacipran (100-200 mg/day dosed twice a day) for radicular pain associated with lumbosacral disk disease.

Outcome measures and safety assessments will be obtained at weeks 1, 2, 4, 6, 8, and 10 according to the protocol schedule of assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female adult outpatient age 18 or older at the time of consent.
2. Subject experiences chronic (> 6 months) radicular pain at least 5 days a week described as sharp or shooting below the level of the knee associated with lumbar or sacral disk disease without suspicion of recent injury; remote (>1 year ago) history of surgical intervention (e.g. "failed back syndrome") is allowed provided current symptoms meet severity criterion.
3. Subject-rated VAS specifically related to radicular pain > or = 40 mm at screen and baseline visits
4. Subject has an understanding, ability and willingness to fully comply with study procedures and restrictions.
5. Subject has the ability to provide written, personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related procedures.

Exclusion Criteria:

1. Subjects unable to complete assessments due to language or cognitive impairment
2. Subjects treated with antidepressant or anticonvulsant medication within 4 weeks of screening visit (6 weeks for fluoxetine).
3. Subjects taking monoamine oxidase inhibitors
4. Subjects who have received procedural intervention within 3 months of screen.
5. Subjects with known sensitivity to milnacipran.
6. Subjects unable to complete the questionnaires due to language or cognitive impairment.
7. Subjects with a history of bipolar disorder or psychosis as confirmed by the Mini International Neuropsychiatric Interview (MINI).
8. Subject currently has (or had a history within the last 6 months of) a drug dependence or substance abuse disorder according to Diagnostic and Statistical Manual for Mental Disorders, Text Revision criteria (excluding nicotine).
9. Subjects who are currently considered a suicide risk, any subject who has previously made a suicide attempt or who has a prior history of or are currently demonstrating active suicidal ideation.
10. Subject has any clinically significant electrocardiogram (ECG) or clinically significant laboratory abnormality (including a positive urine drug screen) at Screening.
11. Subject has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that in the Investigator's opinion would prohibit the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol.
12. Subjects who are pregnant or who are nursing
13. Subjects who do not agree to use adequate and reliable contraception throughout the study.
14. Subject previously completed, discontinued or was withdrawn from this study.
15. Subject has taken an investigational drug or taken part in a clinical trial within 30 days prior to Screening.
16. Subjects with liver disease or reduced liver function
17. Subjects with obstructive uropathies
18. Subjects who consume alcohol in amounts viewed by the Investigator to be contraindicated
19. Subjects with uncontrolled narrow angle glaucoma
20. Subjects with seizure disorders
21. Subjects with bleeding disorders or use of other medications that may cause bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

REFERENCES:
- [Derived] Marks DM, Pae CU, Patkar AA. A double-blind, placebo-controlled, parallel-group pilot study of milnacipran for chronic radicular pain (sciatica) associated with lumbosacral disc disease. Prim Care Companion CNS Disord. 2014 Aug 14;16(4):10.4088/PCC.14m01658. doi: 10.4088/PCC.14m01658. eCollection 2014. PMID 25664215

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Started | 8 (Includes one subject screened/consented but not assigned to either arm.) | 5 (Includes one subject screened/consented but not assigned to either arm.)
Completed | 5 | 3
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two subjects were screened/consented but not assigned to either arm patient. These two patients are reflected as one that would have been assigned to each arm. These subjects were did not receive inerventons
Groups:
- Milnacipran: Milnacipran, flexibly dosed 100-200 mg/day dosed twice a day
- Total: Total of all reporting groups
Arm/Group | Milnacipran | Sugar Pill (Placebo) | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale Score Referring to Radicular Pain (VAS-rad)
Description: The primary outcome is change in pain VAS from baseline through 10 weeks. The effect size was calculated using the VAS scores measured on a scale of 0 to 100 mm with 0 being absence of pain or no pain noted and 100 being worst imaginable pain/as bad as can be. The higher the score the greater the over all pain intensity. Mean cumulative total scores were reported.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Milnacipran: Milnacipran, flexibly dosed (100-200 mg/day dosed twice a day)
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 5 | 3
units on a scale
  Values at baseline | 58.7 (9.4) | 67.7 (26.5)
  Values at endpoint | 13.6 (8.5) | 59.7 (43.6)

2. Secondary Outcome: VAS Related to Nociceptive Pain Component (VAS-Noc)
Description: The secondary outcome is change in pain VAS from baseline through 1o weeks as related to nociceptive pain component. The effect size was calculated using the VAS scores measured on a scale of 0 to 100 mm with 0 being absence of pain or no pain noted and 100 being worst imaginable pain/as bad as can be. The higher the score the greater the over all pain intensity. Mean cumulative scores were reported
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 5 | 3
units on a scale
  Values at baseline | 57.3 (17.2) | 64.7 (43.0)
  Values at endpoint | 32.2 (30.4) | 64.7 (46.3)

3. Secondary Outcome: SF-36 (Short Form)
Description: Self-report of quality of life. Subjective measure of perceived quality of life.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section.
  Scoring: Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Higher scores reflect higher quality of life with 100 high life quality. Total mean cumulative scores were reported
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 5 | 3
units on a scale
  Values at baseline | 96.9 (6.3) | 101.3 (4.0)
  Values at endpoint | 97.0 (5.8) | 99.7 (8.9)

4. Secondary Outcome: Oswestry Low Back Pain Disability Questionnaire
Description: Self report evaluation of various back pain symptoms. For each of 10 sections participants rate pain on a scale of 0-5 in these categories:
  * Section 1 - Pain intensity
  * Section 2 - Personal care
  * Section 3 - Lifting
  * Section 4 - Walking
  * Section 5 - Sitting
  * Section 6 - Standing
  * Section 7 - Sleeping
  * Section 8 - Sex life (if applicable)
  * Section 9 - Social life
  * Section 10 - Travelling
  The scores are combined form each category into overall score. Scores are converted to percentages as follows:
  0% to 20%: minimal disability: The patient can cope with most living activities.
  21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing.
  41%-60%: severe disability: Pain remains the main problem-activities of daily living are affected.
  61%-80%: crippled: Back pain impinges on all aspects of life.
  81%-100%: Patients are either bed-bound or exaggerating their symptoms
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: percent score
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 5 | 3
percent score
  Values at baseline | 20.1 (7.4) | 22.8 (11.2)
  Values at endpoint | 18.1 (8.0) | 22.5 (15.0)

5. Secondary Outcome: Neuropathic Pain Questionnaire
Description: Self-report evaluation of nerve pain symptoms. A low total cumulative score means less pain and higher cumulative score is greater pain.
  Total cumulative scores range form 0 to 1000 where in 0 is absence of pain and 1000 highest pain.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 7 | 4
units on a scale
  Values at baseline | 415.1 (202) | 601.4 (336.7)
  Values at endpoint | 238.3 (279.9) | 511.3 (414.1)

6. Secondary Outcome: Beck Depression Inventory (BDI-II)
Description: Self-report evaluation of depressive symptoms.The secondary outcome measure is change in Beck Depression Inventory. The scale for this inventory is:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. The higher the score the degree of depression.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 5 | 3
units on a scale
  Values at baseline | 13.8 (7.3) | 14.3 (9.3)
  Values at endpoint | 11.6 (8.2) | 13.3 (10.3)

7. Secondary Outcome: State-trait Anxiety Inventory (STAI)
Description: Self-report evaluation of anxiety symptoms.Assessment of subjective symptoms of current anxiety and chronic anxiety.
  There are 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale
  Scale
  1= almost never 4= almost always
  Higher scores indicate greater anxiety. Mean cumulative scores were reported
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Number analyzed (Participants) | 7 | 4
units on a scale
  Values at baseline | 88.4 (7.1) | 86.5 (5.9)
  Values at endpoint | 90.0 (7.9) | 84.0 (10.9)

ADVERSE EVENTS:
Arm/Group | Milnacipran | Sugar Pill (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No